CLINICAL TRIAL: NCT03931330
Title: Does Improving Vagal Tone Increase Mitochondrial Bioenergetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Chelimsky, Gisela Grotewold, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1101710
Record Dates: First submitted 2019-04-22; First posted 2019-04-30 (Actual); Results first posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-05

CONDITIONS: Functional Gastrointestinal Disorders; Irritable Bowel Syndrome; Dyspepsia; Functional Abdominal Pain Syndrome
Keywords: FGID; Neural Stimulation; Functional Abdominal Pain; Dysautonomia
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome; Dyspepsia; Autonomic Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: All subjects will receive the same electro auricular device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Percutaneous neurostimulation (Experimental): Subjects will have 4 weeks of active therapy.
  Interventions: Device: Percutaneous neurostimulation

INTERVENTIONS:
Device: Percutaneous neurostimulation — Percutaneous neurostimulation using NSS-2 Bridge device
  Other Names: NSS-2 Bridge by Innovative Health Solutions

SUMMARY:
This study evaluates the effect of auricular neurostimulation on mitochondrial bioenergetics and inflammation through vagal nerve modulation via non-invasive percutaneous electrical nerve field stimulator in children with functional gastrointestinal disorders.

DETAILED DESCRIPTION:
In understanding the pathophysiology of pediatric functional gastrointestinal disorders (FGID), it has been documented that subjects have decreased vagal tone. Vagal tone in turn modulates mitochondrial bioenergetics and plays a role in anti inflammatory effects. Further defining these brain-body connections that underlie FGID's could help guide future treatment.

The investigators postulate that a 4 week neuro-stimulation with an Electro Auricular Device that has already shown to increase vagal tone will produce an increase in mitochondrial bioenergetics and decrease in inflammatory markers in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking and able to verbalize their condition and concerns about nausea, pain and other symptoms
* Subjects will meet Rome IV criteria for functional nausea, irritable bowel syndrome, dyspepsia or functional abdominal pain as determined by a pediatric gastroenterologist
* Patients must have an intact external ear that is free of infection or severe dermatological conditions, have stable vital signs for their respective age, no history of seizures and no currently implanted electrical device

Exclusion Criteria:

* Mental retardation or pervasive developmental disorder or epilepsy
* Psychosis
* Genetic or chromosomal disorders
* Pregnancy
* Subjects who admit to substance abuse during screening
* Patients with findings of peptic ulcer disease, H.pylori gastritis, celiac disease, inflammatory bowel disease, allergic disorders, or any chronic condition or medication that may cause nausea or pain
* Patients who are treated with opioids or who had any changes in their medical regimen in the past four weeks prior to study
* Patients with a history of allergy to adhesives

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Chelimsky, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He X, Zhao M, Bi X, Sun L, Yu X, Zhao M, Zang W. Novel strategies and underlying protective mechanisms of modulation of vagal activity in cardiovascular diseases. Br J Pharmacol. 2015 Dec;172(23):5489-500. doi: 10.1111/bph.13010. Epub 2015 Jan 13. PMID 25378088
- [Background] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627
- [Background] Liu Q, Wang EM, Yan XJ, Chen SL. Autonomic functioning in irritable bowel syndrome measured by heart rate variability: a meta-analysis. J Dig Dis. 2013 Dec;14(12):638-46. doi: 10.1111/1751-2980.12092. PMID 23927739

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited form the pediatric neurogastrointestinal clinic, from 2/6/2019 to 5/23/2019
Groups:
- Only Active Devise, Open Label: active devise, 4 weeks
Period: Overall Study
Arm/Group | Only Active Devise, Open Label
Started | 8
4 Weeks of Neuromodulation | 7 (at 4 weeks of neuromodulation)
Completed | 7
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Percutaneous Neurostimulation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: To Measure Different Mitochondrial Bioenergetic Markers, Including Basal Respiratory Capacity
Description: Blood draw will be tested for mitochondrial function, including basal respiratory capacity, ATP production and spare respiration and to detect changes in protein which can be an indicator for inflammation. Basal Respiratory Capacity (pmol/min) is better when value is higher.
Time Frame: Baseline, at follow-up visit 4 (Week 4) and at follow up visit 5 (Week 8 or 12)
Population: Per protocol maximal respiration data was collected for patients at baseline, after completing all 4 weeks of NSS Bridge Neurostim therapy and long term follow up post therapy.
Measure: Mean (Standard Deviation); unit: pmol/min
Groups:
- Only Active Devise, Open Label: Mitochondrial bioenergetics is decreased in adolescents with FGID, we postulate that a 4 week neuro-stimulation with an EAD that has already shown to increase vagal tone will produce an increase in mitochondrial bioenergetics in this patient group.
Arm/Group | Only Active Devise, Open Label
Number analyzed (Participants) | 7
pmol/min
  Week 1 | 221.85 (195.35)
  Week 4 | 151.14 (101.97)
  Week 8 | 139.20 (120.12)

2. Secondary Outcome: To Measure Heart Rate Variability
Description: EKG tracing will be used to analyze Heart Rate Variability as an indirect measure of vagal nerve output and central autonomic control.
Time Frame: At date of baseline assessment (beginning of therapy). Also assessed at follow-up visit 4 (Week 4) and 5 (Week 8 or 12)
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Only Active Devise, Open Label
Number analyzed (Participants) | 7
Beats per minute
  Week 1 | 100.31 (17.31)
  Week 4 | 97.27 (21.69)
  Week 8 | 93.86 (15.63)
  Total | 97.35 (18.17)

3. Secondary Outcome: To Measure Functional Disability Inventory
Description: The Functional Disability Inventory (FDI) questionnaire will be used to assess change in symptoms. Participants will rank physical trouble or difficulty completing 15 different daily activities (Eating regular meals, Being at school all day, Walking up stairs, etc.) on a scale of 0-4.
  Scale:0-No trouble
  1. A little trouble
  2. Some Trouble
  3. A lot of Trouble
  4. Impossible
  Higher scores (4) indicate more difficulty functioning due to physical health. The total score ranges from 0 to 60 among 15 questions. The individual score for all 15 questions are added together for the total score. If all 15 questions are answered as 0- no trouble then the total score would be 0 (lowest difficulty). If all 15 questions are answered as 4-Impossible, then the total score would be 60 (highest difficulty). An assortment of answers will fall within this 0-60 range depending on the difficulty level answer for each question.
Time Frame: At date of baseline assessment (beginning of therapy). Also assessed at follow-up visit 4 (Week 4) and visit 5 (8 or 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Only Active Devise, Open Label
Number analyzed (Participants) | 7
score on a scale
  Week 1 | 26.53 (14.04)
  Week 4 | 24.58 (15.25)
  Week 8 | 22.70 (17.47)
  Total | 24.74 (14.60)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 weeks, including the follow up visit
Groups:
- Only Active Device, Open Label: active device, 4 weeks
Arm/Group | Only Active Device, Open Label
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT03931330/Prot_SAP_000.pdf